CLINICAL TRIAL: NCT02156869
Title: Impact of a Printed Decision Aid on Patients' Intent to Undertake Prostate Cancer Screening: a Multicenter Pragmatic Randomized Controlled Trial
Brief Title: Impact of a Printed Decision Aid on Patients' Intent to Undertake Prostate Cancer Screening
Acronym: PSAMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, TRAN Viet thi, Assistant professor, University Paris 7 - Denis Diderot
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DMG1
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Screening; Decision aids
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): The intervention was the use of a decision aid.
  Interventions: Other: Decision aid
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Other: Decision aid — Intervention was use of a decision aid. Decision aid contained information about: 1) the epidemiology of prostate cancer; 2) what is a PSA test and advantages and limits of screening for prostate cancer using it (including risk of overtreatment and risk of becoming impotent and/or incontinent) and; 3) the position on screening for prostate cancer of major scientific societies in France at the time of the study. The second page contained a visual representation of the benefits of PSA screening for prostate cancer versus usual care based on the results of the European Randomized study of Screening for Prostate Cancer trial (ERSPC) The decision aid was pretested with 20 patients to ensure clarity and wording. It was revised accordingly to comments.
  Arms: Intervention arm

SUMMARY:
Although the number of recommendations against systematic screening of prostate cancer, 70% of patients still request testing because they overestimate the benefits and are unaware of the limitations.

The investigators aim is to assess the impact of a short printed decision aid presenting benefits and limits of screening, on patients' intent to undergo prostate cancer screening.

DETAILED DESCRIPTION:
A Cochrane systematic review of 5 randomized controlled trials showed that screening for prostate cancer, using digital rectal examination and dosage of prostate specific antigen (PSA), did not significantly decrease prostate cancer specific mortality. Rather, screening for prostate cancer often led to over-diagnosis by detecting tumors that would not otherwise have become symptomatic or by producing false positive results. It could therefore result in unnecessary supplementary testing (including prostate biopsies), inadequate and/or harmful treatment, and negative psychological outcomes among patients.

Although the growing number of recommendations against PSA testing for screening of prostate cancer, 70% of patients still request testing prior to any information because they overestimate the benefits and are unaware of the limitations. As a result, about 55% of patients between 50 and 74 years old, undergo prostate cancer screening in the USA every year, despite recommendations against it.

To help patients understand the complexities about PSA testing for prostate cancer screening, professional organizations encourage physicians and patients to use decision aids to make informed decisions.

The aim of this study was to evaluate the impact of a decision aid, usable in daily practice by general practitioners, presenting harms and benefits of prostate cancer screening on patients' intent to undergo screening.

ELIGIBILITY:
Inclusion Criteria:

* male patients from 50 to 75 years old

Exclusion Criteria:

* personal history of prostate cancer
* any urinary tract symptoms
* history of prostate cancer in a first degree relative
* known exposition to chlordecone

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
patients' intent to undergo screening for prostate cancer | Immediate
  patients' intent to undergo screening for prostate cancer was assessed by the question: "Do you want to be screened (or in case you have already been screened before, do intend to continue to be screened) for prostate cancer?" in a self administered questionnaire. Patients could answer "Yes", "No" or "I don't know", measured one time after receiving the decision aid or not.

OTHER OUTCOMES:
Reasons to undergo or not screening for prostate cancer | Immediate
  We systematically asked patients to elicit reasons underlying their answers using open-ended questions. Answers were read by a single investigator (EKR) and classified into categories. We compared proportion of individuals eliciting ech reason between the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: Viet Thi Tran, MD, Principal Investigator — Paris Diderot University
Locations (1):
- SFTG, Paris, France

REFERENCES:
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for prostate cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Jul 17;157(2):120-34. doi: 10.7326/0003-4819-157-2-201207170-00459. PMID 22801674
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076